CLINICAL TRIAL: NCT00259168
Title: Insulin Resistance and Postprandial Endothelial Function: Does Early Intervention Make a Difference?
Brief Title: Insulin Resistance and Vessel Function After Meals: Does Early Intervention Make a Difference?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Atheline Major-Pedersen (Other)
Collaborators: Novartis (Industry); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Atheline Major-Pedersen, MD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-005/03
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Insulin Resistance; Impaired Fasting Glucose
Keywords: Postprandial endothelial function
MeSH Terms: conditions — Insulin Resistance | interventions — Nateglinide

INTERVENTIONS:
Drug: Nateglinide

SUMMARY:
The purpose of this study is to determine whether attenuation/normalization of elevated blood sugar after meals ameliorates vessel wall (endothelial) function in individuals with insulin resistance.

DETAILED DESCRIPTION:
Background:Insulin Resistance (IR) is accompanied by a high incidence and prevalence of cardiovascular disease. IR is present in individuals with pre-diabetes/ type 2 diabetes. Epidemiological data demonstrate a tight relationship between postprandial blood sugar, insulin resistance and cardiovascular disease (CVD). Endothelial dysfunction seems to be the very first sign of CVD.

Purpose: We propose to determine whether attenuation /normalization of post-prandial hyperglycaemia, through the administration of an oral hypoglycaemic agent of ultra rapid action (nateglinide), ameliorates endothelial function in the IR.

We extrapolate that a better endothelial function in the brachial artery reflects regression of atherosclerotic changes in the coronary system.

Method and Study Design: Prospective, open, parallel, group comparison study of 1 intervention group, 1 intervention control group and 1 disease control group. The intervention group and the intervention control group each consist of 30 individuals with IR. Individuals in the intervention group receive an individually adjusted dose of nateglinide 3 times daily during 12 weeks. The third group consists of 10 healthy, young individuals. All groups are followed during 3 months with an otherwise unchanged lifestyle. Endothelial function is measured with the Flow Mediated Dilation method before and after the intervention/observation period.

ELIGIBILITY:
Inclusion Criteria:

* Insulin resistance, impaired glucose tolerance

Exclusion Criteria:

* unstable chronic disease, acute disease

Ages: 25 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Endothelial function

SECONDARY OUTCOMES:
Metabolic function

CONTACTS AND LOCATIONS:
Overall Officials: Christian Torp-Pedersen, MD, DMSc, Study Chair — Bispebjerg Hospital
Locations (1):
- Endothelial laboratory, Cardiology clinic Y-research, H:S Bispebjerg Hospital, Bispebjerg Bakke, Copenhagen, Copenhagen NV, Denmark

REFERENCES:
- [Background] Ceriello A, Taboga C, Tonutti L, Quagliaro L, Piconi L, Bais B, Da Ros R, Motz E. Evidence for an independent and cumulative effect of postprandial hypertriglyceridemia and hyperglycemia on endothelial dysfunction and oxidative stress generation: effects of short- and long-term simvastatin treatment. Circulation. 2002 Sep 3;106(10):1211-8. doi: 10.1161/01.cir.0000027569.76671.a8. PMID 12208795
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217